CLINICAL TRIAL: NCT02634606
Title: Effects of a Tocotrienol-Enriched Fraction of Palm Oil on Serum Lipids in Hypercholesterolemic Subjects
Brief Title: Effects of a Supplement Derived From Palm Oil on Cholesterol Levels in the Blood
Acronym: TRF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to obtain supplement for this study. Unable to recruit.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: TOCO 11-000665
Record Dates: First submitted 2014-09-26; First posted 2015-12-18 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gamma Delta Tocotrienols - Low Dose (Active Comparator): 33 subjects with cholesterol level (>180 mg/dl), ages 35-70, currently taking statins who meet all of the eligibility criteria in the screening phase of the study will be assigned to the TRF (63mg) arm of the study to evaluate the cholesterol suppressive actions of TRF. Subjects will be asked to take 2 tablets per day and to maintain the American Heart Association (AHA) diet for 12 weeks.
  Interventions: Drug: Gamma Delta Tocotrienols - Low Dose
- Gamma Delta Tocotrienols - High Dose (Active Comparator): 33 subjects with cholesterol level (>180 mg/dl), ages 35-70, currently taking statins who meet all of the eligibility criteria in the screening phase of the study will be assigned to the TRF (127mg) arm of the study to evaluate the cholesterol suppressive actions of TRF. Subjects will be asked to take 2 tablets per day and to maintain the American Heart Association (AHA) diet for 12 weeks.
  Interventions: Drug: Gamma Delta Tocotrienols - High Dose
- Sugar Pill (Placebo Comparator): 33 subjects with cholesterol level (>180 mg/dl), ages 35-70, currently taking statins who meet all of the eligibility criteria in the screening phase of the study will be assigned to the Placebo arm of the study to evaluate the cholesterol suppressive actions of Placebo. Subjects will be asked to take 2 tablets per day and to maintain the American Heart Association (AHA) diet for 12 weeks.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Gamma Delta Tocotrienols - Low Dose — 250 mg capsule containing 63 mg Gamma Delta Tocotrienols 2x/day for 12 weeks.
  Other Names: Tocotrienol-enriched Fraction of Palm Oil (TRF)
  Arms: Gamma Delta Tocotrienols - Low Dose
Drug: Gamma Delta Tocotrienols - High Dose — 250 mg capsule containing 127 mg Gamma Delta Tocotrienols 2x/day for 12 weeks.
  Other Names: Tocotrienol-enriched Fraction of Palm Oil (TRF)
  Arms: Gamma Delta Tocotrienols - High Dose
Drug: Sugar Pill — 250 mg Placebo capsule containing 50% medium chain triglycerides and 50% glycerin 2x/day for 12 weeks.
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
Elevated blood cholesterol, and particularly LDL cholesterol, is a risk factor for heart disease. Tocotrienols are naturally-occurring compounds in foods that may have beneficial effects on blood cholesterol. Tocotrienols are members of the vitamin E family, and are found in barley, oats, rye, coconut oil and rice bran oil, but the richest source of tocotrienols is palm oil. Certain of these tocotrienols have been shown to be effective in lowering LDL (or 'bad') cholesterol, with no adverse effects on the HDL (or 'good') cholesterol. The purpose of this study is to determine the effects of a palm-oil derived tocotrienol supplement on blood cholesterol, and particularly LDL cholesterol, in individuals who are taking statins, and have either elevated or normal cholesterol levels. Study subjects will consume a palm-oil derived supplement of tocotrienol for 3 months to determine its effects on LDL cholesterol.

DETAILED DESCRIPTION:
Both tocotrienols and tocopherols, whose derivatives are in eight different isoforms, are closely related structurally. Tocopherols are generally present in common vegetable oils (i.e. soy, canola). However, tocotrienols are concentrated in cereal grains (ie. oat, barley, and rye, rice bran), with the highest level found in crude palm oil. The development of new cholesterol-lowering agents has been given more and more attention by pharmaceutical companies due to the strong relationship between cholesterol and atherosclerosis. Tocotrienols, especially δ- and γ-tocotrienols, were shown to be effective nutritional agents to treat high cholesterol in recent research programs. In particular, γ-tocotrienol appears to inhibit 3-hydroxy-3-methylglutaryl-coenzyme A reductase at a posttranscriptional level and there is some evidence that tocopherols antagonize this effect. Therefore, the current study is designed to demonstrate that treatment with a tocotrienol-enriched fraction of palm oil for a three month period will lead to a significant reduction in LDL cholesterol with no effect on HDL cholesterol in patients whose cholesterol level is not adequately controlled in spite of statins. This objective will be achieved utilizing a simple three arm randomized placebo-controlled trial in a total of 99 subjects After acclimation to a step I AHA diet and no supplemental vitamin E in the diet, subjects will be given either a placebo capsule or a tocotrienol (120mg or 240mg) capsule in addition to their statin medications

ELIGIBILITY:
Inclusion Criteria:

* Able to read, speak, and understand English
* Male or female, 35-70 years old (inclusive)
* Total Fasting Plasma Cholesterol of >180 mg/dl
* Currently taking statin medications.
* Willing to maintain AHA Step 1 diet for the duration of the study.

Exclusion Criteria:

* Any subject who is taking vitamin E supplements or taking any antibiotics or other medication or dietary supplement which could interfere with the action of tocotrienols.
* Any subject who is taking cholesterol lowering medications other than statins.
* Any subject who has lost >5% of their body weight during the past 3 months.
* Any subjects with a history of gastrointestinal surgery, diabetes mellitus, or other serious medical condition, such as chronic hepatitis or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as BP >160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
* Major surgery within 12 weeks prior to subject randomization and/or screening, especially cardiac surgery
* Is currently a smoker who has a therapeutic plan to quit smoking anytime during the study period; or if not a current smoker, has quit smoking within the past 3 months.
* Known HIV positive or known immunocompromised condition (e.g. MV, organ transplantation, treatment with immunosuppressant medications).
* Clinical evidence of current malignancy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia.
* Currently receiving systemic chemotherapy and/or radiotherapy.
* Active bleeding.
* Subject has any disorder (excluding illiteracy or visual impairment) that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
* In the opinion of the study investigator has a risk of non-compliance with study procedures, or cannot read, understand or complete study related materials.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2015-11-13 (Actual); Study Completion 2015-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles; David Heber, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, 900 Veteran Avenue, WH 14-187, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 3/22/2011 - 11/13/2015 and took place in a private setting the clinic located at the site.
Pre-assignment Details: Thirteen subjects with cholesterol level (>180 mg/dl), aged 37-64, taking statins drug at the time were to be assigned to the low dose arm (TRF 63 mg), high dose arm (RTF 127 mg) or control (sugar pill) for 12 weeks. Randomization was not performed due to limited subjects recruited.
Groups:
- Pre-Randomization: Thirteen enrolled subjects were to be assigned to the low dose arm (TRF 63 mg), high dose arm (RTF 127 mg) or control (sugar pill). Randomization was not performed prior to study termination.
Period: Overall Study
Arm/Group | Pre-Randomization
Started (13 eligible participants enrolled; none were assigned to an intervention prior to termination.) | 13
Completed | 0
Not Completed | 13
Not completed — unable to obtain the drug at start | 13

BASELINE CHARACTERISTICS:
Population: Enrolled subjects were not assigned to an intervention arm prior to study termination.
Arm/Group | Pre-Randomization
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in LDL Cholesterol Over Time Between the 3 Groups
Description: Mixed-effects regression models will be used to evaluate the change in LDL cholesterol over time between the 3 groups
Time Frame: Baseline and 12 weeks
Population: Randomization was not performed prior to study termination
Arm/Group | Gamma Delta Tocotrienols - Low Dose | Gamma Delta Tocotrienols - High Dose | Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not reported/collected because no participants were assigned to an intervention arm prior to study termination
Arm/Group | Gamma Delta Tocotrienols - Low Dose | Gamma Delta Tocotrienols - High Dose | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No